CLINICAL TRIAL: NCT01386931
Title: The Clinical Impact of Immediate On-site Cytopathology Evaluation During Endoscopic Ultrasound-Guided Fine Needle Aspiration of Pancreatic Mass: A Multicenter, Prospective Randomized Controlled Trial
Brief Title: On-site Cytopathology EUS-FNA
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 11-0919; 11-0919 (Other: Siteman Cancer Center PRMC)
Record Dates: First submitted 2011-06-27; First posted 2011-07-01 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Pancreatic Neoplasms; Pancreatic Cancer
Keywords: Biopsy, Fine-Needle; Endoscopic Ultrasonography; cytopathology
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cytopathologist present during EUS-FNA: Patients assigned to the on-site cytopathologist arm will have the cytopathologist dictate the number of FNA passes performed by the endosonographer. This number will be based on the adequacy of specimen and the ability to provide a preliminary diagnosis.
  After EUS-FNA is performed all slides will be sent to the pathology department. The slides will be sent for review regardless of which arm the patient is randomized into, and they will be reviewed by experienced cytopathologists for the purpose of determining the final diagnoses.
  Interventions: Procedure: EUS-guided FNA performed with on-site Cytopathologist
- Cytopathologist absent during EUS-FNA: In the absence of an on-site cytopathologist, the endosonographer will perform a predetermined number of 7 passes (standard of care in the absence of an on-site cytopathologist).
  After EUS-FNA is performed all slides will be sent to the pathology department. The slides will be sent for review regardless of which arm the patient is randomized into, and they will be reviewed by experienced cytopathologists for the purpose of determining the final diagnoses.
  Interventions: Procedure: EUS-guided FNA performed without on-site Cytopathologist

INTERVENTIONS:
Procedure: EUS-guided FNA performed with on-site Cytopathologist — Patients assigned to the on-site cytopathologist arm will have the cytopathologist dictate the number of FNA passes performed by the endosonographer. This number will be based on the adequacy of specimen and the ability to provide a preliminary diagnosis.
  Groups: Cytopathologist present during EUS-FNA
Procedure: EUS-guided FNA performed without on-site Cytopathologist — In the absence of an on-site cytopathologist, the endosonographer will perform a predetermined number of 7 passes (standard of care in the absence of an on-site cytopathologist).
  Groups: Cytopathologist absent during EUS-FNA

SUMMARY:
This study is a multicenter prospective randomized controlled trial. Potential participants in this study include patients referred for Endoscopic Ultrasound-guided fine needle aspiration (EUS-FNA) of a solid pancreatic lesion at one of the participating centers. If the patient meets inclusion criteria and signs the informed consent, they will be randomized into one of the two study arms in a 1:1 ratio. Patients will either undergo EUS-FNA with or without an on-site cytopathologist present during EUS-FNA. Patients assigned to the on-site cytopathologist arm will have the cytopathologist dictate the number of fine needle aspiration (FNA) passes performed by the endosonographer. This number will be based on the adequacy of specimen and the ability to provide a preliminary diagnosis. In the other arm, in the absence of an on-site cytopathologist, the endosonographer will perform a predetermined number of 7 passes (standard of care in the absence of an on-site cytopathologist). The technique of performing EUS-FNA (needle type, use of stylet, suction) will be standardized among all endosonographers in order to rule out confounding factors. After EUS-FNA is performed all slides will be sent to the pathology department. The slides will be sent for review regardless of which arm the patient is randomized into, and they will be reviewed by experienced cytopathologists for the purpose of determining the final diagnoses.

Future clinical intervention will be monitored for the purpose of reporting the impact EUS-FNA has on the patient's clinical course and determining diagnostic accuracy. Patients will be followed prospectively for at least one year, and the gold-standard for final diagnosis of pancreatic malignancy will be defined by the presence of malignant cytology or histologic evidence (if the patient undergoes surgery) or with clinical and/or imaging follow-up consistent with pancreatic cancer (death or clinical progression). A detailed account of medical equipment used during each procedure, procedure time, clinic visits/hospitalizations due to procedure related complications, and number of repeat procedures will be recorded systematically.

The investigators hypothesize that an on-site cytopathologist during EUS-FNA for pancreatic masses improves diagnostic yield, accuracy, and lowers the duration, complications and the need for repeat procedures.

DETAILED DESCRIPTION:
Endoscopic Ultrasound (EUS) plays an integral role in the diagnosis of suspected pancreatic cancer, and the EUS findings are crucial for determining the course of future management and potential treatment options for these patients. EUS is the most sensitive imaging modality for the detection of pancreatic masses, and has a sensitivity of greater than or equal to 90%. Furthermore, EUS-guided fine needle aspiration (EUS-FNA) plays an important role in accurate staging of pancreatic cancer with a sensitivity of 85% and specificity close to 100%. EUS-FNA is considered to be cost-effective by virtue of its impact on therapeutic management. In particular, real-time tissue sampling by EUS-FNA is possible when a cytopathologist (pathologist skilled in evaluating fine needle aspiration specimens) is able to be present at the time of FNA in order to review the biopsy slides and make a preliminary diagnosis. The availability of an on-site cytopathologist has the potential to provide quick diagnostic and predictive information to confirm the presence and staging of suspected malignancy. The rationale for an on-site cytopathologist includes increasing the adequacy and yield of biopsy tissue/aspirate which can decrease the need for additional passes to obtain a diagnostic yield of tissue. This hypothesis, however, has not been formally examined.

In this proposed randomized controlled multicenter trial, the investigators hypothesize that an on-site cytopathologist during EUS-FNA for pancreatic masses improves diagnostic yield, accuracy, and lowers the duration, complications and the need for repeat procedures. This hypothesis will be explored in the context of the following specific aims.

Specific aim #1: To compare the diagnostic yield of malignancy and proportion of inadequate specimens between the two groups.

Specific aim #2: To compare the sensitivity, specificity and accuracy of EUS-FNA between the two groups using histologic diagnosis or cytologic diagnosis in conjunction with clinical and/or imaging follow-up as the gold standard.

Specific aim #3: To compare the duration, rate of complications and repeat procedures between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients age: greater than or equal to 18 years
* Presence of a solid pancreatic mass lesion confirmed by at least a single investigational modality such as computerized axial tomography (CT) scan, magnetic resonance imaging (MRI) or Endoscopic Ultrasound (EUS)
* Ability to provide written informed consent

Exclusion Criteria:

* Severe coagulopathy [International Normalized Ratio (INR) > 1.8] or thrombocytopenia (platelet count <50,000)
* Pure cystic lesions of the pancreas
* Inability to sample lesion due to the presence of intervening blood vessels
* Results of EUS-FNA would not impact patient management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants for this study include patients presenting to each of the three tertiary referral centers for an Endoscopic Ultrasound-guided Fine Needle Aspiration.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Compare the percent of patients with a positive diagnosis of malignancy in each of the two groups. | 1 year from the time of patient enrollment
  The Investigators would like to look at each of the two groups to assess whether or not having an onsite cytopathologist during EUS-FNA increases the diagnostic accuracy of pancreatic malignancies. To do this, the Investigators will compare the percent of patients in each group who were accurately diagnosed with a malignancy during EUS-FNA to see if the on-site cytopathologist group yields a higher percent of positively diagnosed malignancies.
Compare the percent of patients with inadequate samples (defined by an absence of cellular elements to account for a mass/lesion) between the two groups | 1-2 weeks from patient enrollment/EUS-FNA
  Final slides will be reviewed by three experienced cytopathologists blinded to the patient's randomization group. The slides for each pass will be assessed for: cellularity, adequacy of specimen, contamination, amount of blood, and diagnosis. Using the cytopathologists' assessment of the FNA specimens, the Investigators will compare the percent of patients with inadequate samples in each group to see if the absence of an on-site cytopathologist corresponds with a higher percent of inadequate FNA samples.

SECONDARY OUTCOMES:
Compare the sensitivity, specificity and accuracy of EUS-FNA between the two groups | 1 year from patient enrollment
  Sensitivity, specificity and accuracy of EUS-FNA will be evaluated using histologic diagnosis or cytologic diagnosis in conjunction with clinical and/or imaging follow-up as the gold standard.
Compare the mean number of passes in the two groups | 1 year (length of time it takes to enroll all patients)
  Once all patients have been enrolled and have undergone EUS-FNA with or without an on-site cytopathologist, the Investigators will be able to compare the mean number of fine needle aspiration passes taken during EUS for patients in each group.
Compare the complication rate in the two groups | 1 year (length of time it takes to enroll all patients)
  The complication rates from the two groups of subjects will be evaluated when all subjects have been enrolled.
Compare the EUS procedure duration in each group | 1 year
  The EUS procedure duration from the two groups of subjects will be evaluated when all subjects have been enrolled.
Compare the percent of patients requiring repeat procedures between the groups | 1 year after the time of patient enrollment
  The investigators will follow patients for one year after enrollment to see if they have had any repeat procedures for the purpose of diagnosing their pancreatic mass.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] Sohn TA, Yeo CJ, Cameron JL, Koniaris L, Kaushal S, Abrams RA, Sauter PK, Coleman J, Hruban RH, Lillemoe KD. Resected adenocarcinoma of the pancreas-616 patients: results, outcomes, and prognostic indicators. J Gastrointest Surg. 2000 Nov-Dec;4(6):567-79. doi: 10.1016/s1091-255x(00)80105-5. PMID 11307091
- [Background] Ngamruengphong S, Li F, Zhou Y, Chak A, Cooper GS, Das A. EUS and survival in patients with pancreatic cancer: a population-based study. Gastrointest Endosc. 2010 Jul;72(1):78-83, 83.e1-2. doi: 10.1016/j.gie.2010.01.072. PMID 20620274
- [Background] Turner BG, Cizginer S, Agarwal D, Yang J, Pitman MB, Brugge WR. Diagnosis of pancreatic neoplasia with EUS and FNA: a report of accuracy. Gastrointest Endosc. 2010 Jan;71(1):91-8. doi: 10.1016/j.gie.2009.06.017. PMID 19846087
- [Background] Mertz HR, Sechopoulos P, Delbeke D, Leach SD. EUS, PET, and CT scanning for evaluation of pancreatic adenocarcinoma. Gastrointest Endosc. 2000 Sep;52(3):367-71. doi: 10.1067/mge.2000.107727. PMID 10968852
- [Background] Hunt GC, Faigel DO. Assessment of EUS for diagnosing, staging, and determining resectability of pancreatic cancer: a review. Gastrointest Endosc. 2002 Feb;55(2):232-7. doi: 10.1067/mge.2002.121342. No abstract available. PMID 11818928
- [Background] DeWitt J, Devereaux B, Chriswell M, McGreevy K, Howard T, Imperiale TF, Ciaccia D, Lane KA, Maglinte D, Kopecky K, LeBlanc J, McHenry L, Madura J, Aisen A, Cramer H, Cummings O, Sherman S. Comparison of endoscopic ultrasonography and multidetector computed tomography for detecting and staging pancreatic cancer. Ann Intern Med. 2004 Nov 16;141(10):753-63. doi: 10.7326/0003-4819-141-10-200411160-00006. PMID 15545675
- [Background] Puli SR, Singh S, Hagedorn CH, Reddy J, Olyaee M. Diagnostic accuracy of EUS for vascular invasion in pancreatic and periampullary cancers: a meta-analysis and systematic review. Gastrointest Endosc. 2007 May;65(6):788-97. doi: 10.1016/j.gie.2006.08.028. Epub 2007 Mar 9. PMID 17350008
- [Background] Faigel DO, Ginsberg GG, Bentz JS, Gupta PK, Smith DB, Kochman ML. Endoscopic ultrasound-guided real-time fine-needle aspiration biopsy of the pancreas in cancer patients with pancreatic lesions. J Clin Oncol. 1997 Apr;15(4):1439-43. doi: 10.1200/JCO.1997.15.4.1439. PMID 9193337
- [Background] Eloubeidi MA, Chen VK, Eltoum IA, Jhala D, Chhieng DC, Jhala N, Vickers SM, Wilcox CM. Endoscopic ultrasound-guided fine needle aspiration biopsy of patients with suspected pancreatic cancer: diagnostic accuracy and acute and 30-day complications. Am J Gastroenterol. 2003 Dec;98(12):2663-8. doi: 10.1111/j.1572-0241.2003.08666.x. PMID 14687813
- [Background] Agarwal B, Abu-Hamda E, Molke KL, Correa AM, Ho L. Endoscopic ultrasound-guided fine needle aspiration and multidetector spiral CT in the diagnosis of pancreatic cancer. Am J Gastroenterol. 2004 May;99(5):844-50. doi: 10.1111/j.1572-0241.2004.04177.x. PMID 15128348
- [Background] Williams DB, Sahai AV, Aabakken L, Penman ID, van Velse A, Webb J, Wilson M, Hoffman BJ, Hawes RH. Endoscopic ultrasound guided fine needle aspiration biopsy: a large single centre experience. Gut. 1999 May;44(5):720-6. doi: 10.1136/gut.44.5.720. PMID 10205212
- [Background] Wallace MB, Kennedy T, Durkalski V, Eloubeidi MA, Etamad R, Matsuda K, Lewin D, Van Velse A, Hennesey W, Hawes RH, Hoffman BJ. Randomized controlled trial of EUS-guided fine needle aspiration techniques for the detection of malignant lymphadenopathy. Gastrointest Endosc. 2001 Oct;54(4):441-7. doi: 10.1067/mge.2001.117764. PMID 11577304
- [Background] Lee JH, Stewart J, Ross WA, Anandasabapathy S, Xiao L, Staerkel G. Blinded prospective comparison of the performance of 22-gauge and 25-gauge needles in endoscopic ultrasound-guided fine needle aspiration of the pancreas and peri-pancreatic lesions. Dig Dis Sci. 2009 Oct;54(10):2274-81. doi: 10.1007/s10620-009-0906-1. Epub 2009 Aug 11. PMID 19669880
- [Background] Siddiqui UD, Rossi F, Rosenthal LS, Padda MS, Murali-Dharan V, Aslanian HR. EUS-guided FNA of solid pancreatic masses: a prospective, randomized trial comparing 22-gauge and 25-gauge needles. Gastrointest Endosc. 2009 Dec;70(6):1093-7. doi: 10.1016/j.gie.2009.05.037. Epub 2009 Jul 28. PMID 19640524
- [Background] LeBlanc JK, Ciaccia D, Al-Assi MT, McGrath K, Imperiale T, Tao LC, Vallery S, DeWitt J, Sherman S, Collins E. Optimal number of EUS-guided fine needle passes needed to obtain a correct diagnosis. Gastrointest Endosc. 2004 Apr;59(4):475-81. doi: 10.1016/s0016-5107(03)02863-3. PMID 15044881
- [Background] Erickson RA, Sayage-Rabie L, Beissner RS. Factors predicting the number of EUS-guided fine-needle passes for diagnosis of pancreatic malignancies. Gastrointest Endosc. 2000 Feb;51(2):184-90. doi: 10.1016/s0016-5107(00)70416-0. PMID 10650262
- [Background] Harewood GC, Wiersema LM, Halling AC, Keeney GL, Salamao DR, Wiersema MJ. Influence of EUS training and pathology interpretation on accuracy of EUS-guided fine needle aspiration of pancreatic masses. Gastrointest Endosc. 2002 May;55(6):669-73. doi: 10.1067/mge.2002.123419. PMID 11979248
- [Background] Chang KJ, Katz KD, Durbin TE, Erickson RA, Butler JA, Lin F, Wuerker RB. Endoscopic ultrasound-guided fine-needle aspiration. Gastrointest Endosc. 1994 Nov-Dec;40(6):694-9. PMID 7859967
- [Background] Klapman JB, Logrono R, Dye CE, Waxman I. Clinical impact of on-site cytopathology interpretation on endoscopic ultrasound-guided fine needle aspiration. Am J Gastroenterol. 2003 Jun;98(6):1289-94. doi: 10.1111/j.1572-0241.2003.07472.x. PMID 12818271
- [Background] Cherian PT, Mohan P, Douiri A, Taniere P, Hejmadi RK, Mahon BS. Role of endoscopic ultrasound-guided fine-needle aspiration in the diagnosis of solid pancreatic and peripancreatic lesions: is onsite cytopathology necessary? HPB (Oxford). 2010 Aug;12(6):389-95. doi: 10.1111/j.1477-2574.2010.00180.x. PMID 20662789
- [Background] Tadic M, Kujundzic M, Stoos-Veic T, Kaic G, Vukelic-Markovic M. Role of repeated endoscopic ultrasound-guided fine needle aspiration in small solid pancreatic masses with previous indeterminate and negative cytological findings. Dig Dis. 2008;26(4):377-82. doi: 10.1159/000177025. Epub 2009 Jan 30. PMID 19188731
- [Background] Vilmann P, Saftoiu A. Endoscopic ultrasound-guided fine needle aspiration biopsy: equipment and technique. J Gastroenterol Hepatol. 2006 Nov;21(11):1646-55. doi: 10.1111/j.1440-1746.2006.04475.x. PMID 16984583
- [Background] Ylagan LR, Edmundowicz S, Kasal K, Walsh D, Lu DW. Endoscopic ultrasound guided fine-needle aspiration cytology of pancreatic carcinoma: a 3-year experience and review of the literature. Cancer. 2002 Dec 25;96(6):362-9. doi: 10.1002/cncr.10759. PMID 12478684
- [Background] Savides TJ, Donohue M, Hunt G, Al-Haddad M, Aslanian H, Ben-Menachem T, Chen VK, Coyle W, Deutsch J, DeWitt J, Dhawan M, Eckardt A, Eloubeidi M, Esker A, Gordon SR, Gress F, Ikenberry S, Joyce AM, Klapman J, Lo S, Maluf-Filho F, Nickl N, Singh V, Wills J, Behling C. EUS-guided FNA diagnostic yield of malignancy in solid pancreatic masses: a benchmark for quality performance measurement. Gastrointest Endosc. 2007 Aug;66(2):277-82. doi: 10.1016/j.gie.2007.01.017. PMID 17643700
- [Background] Wani S, Gupta N, Gaddam S, Singh V, Ulusarac O, Romanas M, Bansal A, Sharma P, Olyaee MS, Rastogi A. A comparative study of endoscopic ultrasound guided fine needle aspiration with and without a stylet. Dig Dis Sci. 2011 Aug;56(8):2409-14. doi: 10.1007/s10620-011-1608-z. Epub 2011 Feb 17. PMID 21327919
- [Background] Rastogi A, Wani S, Gupta N, Singh V, Gaddam S, Reddymasu S, Ulusarac O, Fan F, Romanas M, Dennis KL, Sharma P, Bansal A, Oropeza-Vail M, Olyaee M. A prospective, single-blind, randomized, controlled trial of EUS-guided FNA with and without a stylet. Gastrointest Endosc. 2011 Jul;74(1):58-64. doi: 10.1016/j.gie.2011.02.015. Epub 2011 Apr 23. PMID 21514932
- [Derived] Mohamadnejad M, Mullady D, Early DS, Collins B, Marshall C, Sams S, Yen R, Rizeq M, Romanas M, Nawaz S, Ulusarac O, Hollander T, Wilson RH, Simon VC, Kushnir V, Amateau SK, Brauer BC, Gaddam S, Azar RR, Komanduri S, Shah R, Das A, Edmundowicz S, Muthusamy VR, Rastogi A, Wani S. Increasing Number of Passes Beyond 4 Does Not Increase Sensitivity of Detection of Pancreatic Malignancy by Endoscopic Ultrasound-Guided Fine-Needle Aspiration. Clin Gastroenterol Hepatol. 2017 Jul;15(7):1071-1078.e2. doi: 10.1016/j.cgh.2016.12.018. Epub 2016 Dec 23. PMID 28025154